CLINICAL TRIAL: NCT00803920
Title: CGM Substudy, Addendum 2, of the Following Exenatide LAR Protocol 2993LAR-105: A Randomized, Open-Label, Multicenter, Comparator Controlled Study to Examine the Effects of Exenatide Long-Acting Release on Glucose Control (HbA1c) and Safety in Subjects With Type 2 Diabetes Mellitus Managed With Diet Modification and Exercise and/or Oral Antidiabetic Medications)
Brief Title: Continuous Glucose Monitoring (CGM) in Subjects With Type 2 Diabetes Taking Twice-Daily Exenatide or Once-Weekly Exenatide
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: 03404-06-C
Record Dates: First submitted 2008-12-04; First posted 2008-12-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide twice daily or once weekly; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exenatide
- Exenatide LAR

SUMMARY:
The purpose of this substudy is to obtain CGM data from individuals taking exenatide. The CGM measurements gathered before starting and during treatment with exenatide IR and/or exenatide LAR will help determine the characteristics of glucose control during treatment.

ELIGIBILITY:
Inclusion Criteria:

* participant in Amylin Protocol 2993LAR-105
* at least 16 years of age
* type 2 diabetes being treated with stable regiment of metformin, SU, TZD, combination of metformin/SU, combination metformin/TZD, combination SU/TZD
* A1c 7.1 - 11
* fasting glucose less than 280 at screening
* BMI 25 - 45
* stable body weight 6 months prior to screening
* not pregnant and willing to practice birth control
* physical exam & ECG not clinically significant
* lab values judged not to be clinically significant
* able to understand & sign consent form

Exclusion Criteria:

* clinically significant medical condition as judged by investigator
* drug or alcohol abuse
* previous use of exenatide or any GLP-1 analog
* has used any investigational drug in the past 30 days prior to screening
* is currently using: alpha-glucosidase inhibitor, insulin, drugs that affect GI motility, use of systemic corticosteroids, use of medications with addictive potential, prescription or OTC weight-loss medications
* has donated blood within 60 days of screening, or is planning to donate during the study
* has had major surgery or blood transfusion within 2 months of screening
* has had a surgical procedure that may impact gastric emptying
* has any allergies or hypersensitivity to any component of study treatment
* is an immediate family member of personnel affiliated with the study at the investigative site
* is employed by Amylin, Lilly or Alkermes

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to eighteen subjects at the International Diabetes Center study site will be selected for this substudy in accordance with protocol 2993LAR-105
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Characterize glucose control using periodic CGM in subjects participating in protocol 2993LAR-105 at the International Diabetes Center study site. | 2 week periods of time - 3 times during study:
  Baseline CGM will be performed from Visit 2 to Visit 3 for approximately 14 days followed by a second CGM period from Visit 3 to Visit 6 for approximately 17 days. At Week 28, two weeks after Visit 14 (Week 26), subjects will be instructed to begin CGM and to continue through Visit 20 (Week 30) for Group A subjects or Visit 22 (Week 32) for Group B subjects. At Week 50, two weeks after Visit 28 (Week 48), subjects will be instructed to begin the final CGM period and to continue monitoring until the next study visit at Visit 29 (Week 52)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bergenstal, MD, Principal Investigator — Park Nicollet Institute dba International Diabetes Center; Elinor S Strock, APRN, BC, Principal Investigator — Park Nicollet Institute dba International Diabetes Center; Roger S Mazze, PhD, Principal Investigator — Park Nicollet Institute dba International Diabetes Center
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States